CLINICAL TRIAL: NCT06053281
Title: The Role Of Vitamin D For Therapy Responses On Drug Resistant Epilepsy Through Glial-Cell-Line Derived Neurotrophic Factor (GDNF) And Interleukin 1ß (IL-1 ß) Modulation Pathway
Brief Title: The Role of Vitamin D in Neuroinflammatory on Drug Resistant Epilepsy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: DINA KEUMALA SARI (Other)
Responsible Party: Sponsor-Investigator, DINA KEUMALA SARI, Sponsor-investigator, Universitas Sumatera Utara
Organization: Universitas Sumatera Utara (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USU Neuro Pediatric
Record Dates: First submitted 2023-08-29; First posted 2023-09-25 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Drug Resistant Epilepsy
Keywords: vitamin D; GDNF; interleukin
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Intervention Model Description: Double blind
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Experimental): DRE patients with proved vitamin D deficiency (Serum vitamin D level <30ng/ml). intervention: Daily Cholecalciferol 1000 IU in 24 weeks.
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): DRE patients with proved vitamin D deficiency (Serum vitamin D level <30ng/ml). Interventions: Daily Placebo oral (Manufactured to mimic Cholecalciferol) in 24 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Daily Cholecalciferol 1000 IU in 24 weeks
  Other Names: Vitamin D
  Arms: Vitamin D
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The incident of epilepsy still very high in Indonesia, thus many patients become drug resistant epilepsy. As vitamin D has some anticonvulsant effect, the investigators want to study if an additional dose of vitamin D can help with the therapy responses.

DETAILED DESCRIPTION:
Specifically the investigators want to study about :

1. Correlation between serum vitamin D levels and seizure frequency change after vitamin D treatment
2. Correlation between serum GDNF levels and seizure frequency change after vitamin D treatment
3. Correlation between serum Interleukin-1ß levels and seizure frequency change after vitamin D treatment
4. Responder rate. Percentage of patients change of at least 50% of the seizure frequency
5. Remission rate after vitamin D treatment. Percentage of patients without any seizure (seizure freedom)
6. Effect of vitamin D according to epilepsy type. Responder rate in focal and generalized epilepsy.
7. Effect on Global Assesment of the Severity of Epilepsy (GASE)
8. Effect on Hague Seizure Severity scale (HASS)
9. Effect on Quality of Life in Epilepsy in Children: (QOLCE 55)

ELIGIBILITY:
Inclusion Criteria:

1. Age 1 - 18 years
2. Drug-resistant epilepsy
3. Having at least 6 unprovoked seizures in the previous 3 months
4. No vitamin D treatment in the previous 6 months
5. Medication compliance
6. Agreeing to participate in the study
7. Having a social insurance
8. Parental agreement

Exclusion Criteria:

1. Treatments influencing the metabolism of vitamin D other than anticoagulants (rifamycin, isoniazid, ketoconazole, 5-FU fluorouracil, leucovorin)
2. Known hypersensitivity to vitamin D
3. Lost to follow up

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage change of seizure frequency | 12 and 24 weeks
  Change on number of seizure

SECONDARY OUTCOMES:
Correlation between serum vitamin D levels and seizure frequency change after vitamin D treatment | 12 and 24 weeks
  The vitamin D levels (in ng/mL) of each participant is measured at the beginning and the end of the study and then the investigators calculate the seizure frequency change (in percentage, %)
Correlation between serum GDNF levels and seizure frequency change after vitamin D treatment | 12 and 24 weeks
  The serum GDNF levels (in ng/mL) of each participant is measured at the beginning and the end of the study and then the investigators calculate the seizure frequency change (in percentage, %)
Correlation between serum Interleukin-1ß levels and seizure frequency change after vitamin D treatment | 12 and 24 weeks
  The serum Interleukin-1ß levels (in ng/mL) of each participant is measured at the beginning and the end of the study and then the investigators calculate the seizure frequency change (in percentage, %)
Responder rate | 12 and 24 weeks
  Percentage of patients change at least 50% of the seizure frequency
Remission rate after vitamin D treatment | 12 and 24 weeks
  Percentage of patients without any seizure (seizure freedom)
Effect of vitamin D according to epilepsy type | 12 and 24 weeks
  Responder rate in focal and generalized epilepsy
Effect on Global Assessment of the Severity of Epilepsy (GASE) | 12 and 24 weeks
  Effect on Global Assessment of the Severity of Epilepsy (GASE) will be performed at beginning and the end of the study with 7 point Likert in which options are 1 = Not at all severe, 2 = A little severe, 3 = Somewhat severe, 4 = Moderately severe, 5 = Quite severe, 6 = Very severe, 7 = Extremely severe.
Effect on Hague Seizure Severity scale (HASS) | 12 and 24 weeks
  The Hague Seizure Severity scale (HASS) will be performed at beginning and the end of the study with minimum score = 13 to maximum score = 54, in which the lower score indicates the lowest level of seizure severity
Effect on Quality of Life in Epilepsy in Children: (QOLCE 55) | 12 and 24 weeks
  Effect on Quality of Life in Epilepsy in Children: (QOLCE 55) will be performed at beginning and the end of the study with 5 points in which options are 1 = Poor, 2 = Fair, 3 = Good, 4 = Very good, 5 = Excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Dina K. Sari, SpGK(K), Prof.Dr.dr., Principal Investigator — Universitas Sumatera Utara
Locations (1):
- Faculty of Medicine Universitas Sumatera Utara, Medan, North Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: No